CLINICAL TRIAL: NCT00249743
Title: NIH-NIA SBIR Phase I/II Study: Clinical Evaluation of a Device to Reduce Patient Falls
Brief Title: Clinical Evaluation of a Wireless Monitoring Device to Reduce Falls in the Elderly and Others at High Risk of Falling
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NOCwatch International (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 4R44AG022270-02 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2006-05-29 (Estimated); Status verified 2006-05

CONDITIONS: Accidental Falls; Fractures; Injuries
Keywords: fall prevention; fall risk management; RCT; cost
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries

INTERVENTIONS:
Device: FallSaver (formerly called NOCwatch)

SUMMARY:
Falls are a public health problem of significant social and economic significance. No primary intervention devices have been shown to be effective in reducing falls and associated injuries. The objective of this study was to determine whether the new wireless FallSaver device reduces falls and fall-related injuries in elderly skilled nursing facility (SNF) residents. A randomized, prospective, open-label, cross-over study was conducted over a six-month period. The FallSaver device reduced the frequency of falls by 50% and fall-related injuries by 82% in 43 elderly at-risk SNF residents studied over 4,222 patient-days. The device and associated patch enclosure was well tolerated and devoid of serious problems. Significant cost savings and fewer reductions in quality of life are possible if fall-related injuries can be reduced.

DETAILED DESCRIPTION:
OBJECTIVE. No existing devices have proven effective in preventing falls in at-risk individuals. The objective of this study was to determine whether the FallSaver device reduces falls and fall-related injuries in elderly skilled nursing facility (SNF) residents.

DESIGN. This was a randomized, prospective, open-label, cross-over study conducted over a six-month period.

SETTING: The study took place in a 100-bed State Veterans SNF in Washington State.

PARTICIPANTS. Forty-four subjects with anticipated institutional stays of at least 120 days participated in the study. The subjects' mean age was 82.2 + 7.1 years and all were rated high fall risks using the Morse scale.

INTERVENTION Subjects were randomly assigned to the FallSaver device or no device (Observation) for 60 days. Following the end of the 60-day period subjects were crossed over to the opposite treatment. The device, enclosed in an adhesive patch, was applied to the subject's thigh.

MAIN OUTCOME MEASURE The primary outcome measures were falls and fall-related injuries. Secondary outcomes were falls resulting from documented attempts to stand or ambulate without assistance, skin-tolerance to the patch, and compliance.

RESULTS. Total patient-days for the FallSaver and Observation phases were 1,923 and 2,299, respectively. A total of 37 falls occurred in 18 subjects. Thirteen falls occurred during the FallSaver phase and 24 during Observation (p = < 0.05). A total of 7 fall-related injuries occurred; one during the FallSaver phase and 6 during Observation (p = < 0.01). Nineteen falls resulted from documented attempts to stand or ambulate without assistance, six during the FallSaver phase and 13 during Observation (p = < 0.05). The patch was well tolerated and no serious adverse effects were observed.

CONCLUSION. The FallSaver device reduced the frequency of falls by 50% and fall-related injuries by 82% in elderly at-risk SNF residents. The device and associated patch enclosure was well tolerated and devoid of serious problems. Significant cost savings and fewer reductions in quality of life are possible if fall-related injuries can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Residents of a skilled nursing facility. An anticipated institutional stay of at least 120 days. Individuals with a high risk of falling according to the Morse scale (a score of 55+).

Exclusion Criteria:

* Individuals who were allowed to self-ambulate. Individuals with a history of adverse reactions to medical adhesives. Individuals with a history or presence of significant skin breakdown on the legs.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2004-12; Study Completion 2005-07

PRIMARY OUTCOMES:
Falls and fall-related injuries.

SECONDARY OUTCOMES:
Falls resulting from documented attempts to stand or ambulate without assistance.
Skin tolerance to the adhesive.
Compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E Kelly, DrPH, Study Director — NOCwatch International, Inc.; Dennis Clifton, PharmD, Principal Investigator — Washington State University
Locations (1):
- Spokane Veterans Homes, Spokane, Washington, United States

REFERENCES:
- [Background] Kelly KE, Phillips CL, Cain KC, Polissar NL, Kelly PB. Evaluation of a nonintrusive monitor to reduce falls in nursing home patients. J Am Med Dir Assoc. 2002 Nov-Dec;3(6):377-82. doi: 10.1097/01.JAM.0000036702.12824.82. PMID 12807607